CLINICAL TRIAL: NCT05458401
Title: EUropean Real-world Experience Of Previously Treated Advanced/Metastatic HER2-positive Breast Cancer Patients Accessing Trastuzumab Deruxtecan Through a Named Patient Program (EUROPA T-DXd)
Brief Title: EUropean Real-world Experience Of Previously Treated Advanced/Metastatic HER2-positive Breast Cancer Patients Accessing Trastuzumab Deruxtecan
Acronym: EUROPA T-DXd
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: DS8201-0002-EAP-MA
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: HER2-positive Breast Cancer
Keywords: HER2-positive Breast Cancer; Trastuzumab Deruxtecan
MeSH Terms: interventions — trastuzumab deruxtecan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Trastuzumab Deruxtecan (T-DXd) Cohort: Patients with advanced/metastatic HER2-positive breast cancer who are receiving treatment (or previously treated) with trastuzumab deruxtecan (T-DXd).
  Interventions: Drug: Trastuzumab deruxtecan

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — No drug will be administered during this study.
  Other Names: T-DXd

SUMMARY:
A named patient program (NPP) was initiated to allow patients with an unmet medical need to access trastuzumab deruxtecan (T-DXd) treatment. To gain early insights on the use of T-DXd outside of a trial setting, patients with advanced/metastatic HER2+ breast cancer receiving treatment (or previously treated) with T-DXd through the NPP will be invited to participate.

DETAILED DESCRIPTION:
The antibody-drug conjugate T-DXd has been granted conditional approval in the European Union as a single agent for adult patients with unresectable or metastatic HER2+ breast cancer who have previously received ≥2 HER2-based regimens. This was based on data from the Phase II DESTINY-Breast01 trial (NCT03248492).

DS8201-0002-EAP-MA is a real world data (RWD) observational data collection inviting patients with advanced/metastatic HER2+ breast cancer receiving T-DXd through the NPP already to participate to help further understand the usage in a real world clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Participants for whom T-DXd treatment is indicated, according to the summary of product characteristics conditionally approved by the EMA, that are eligible for treatment with T-DXd through the NPP (i.e., those with advanced/metastatic HER2+ breast cancer who have received ≥ 2 prior anti-HER2-based regimens and have documentation of HER2 positive tumour status by a validated method) will be eligible for inclusion to this RWD collection, subject to providing written informed consent to participate.

Exclusion Criteria:

* Any participant who does not meet all inclusion criteria noted above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The real world data (RWD) collection will include adult participants with advanced/metastatic HER2+ breast cancer treated in routine clinical practice. The collection of RWD will be optional and independent to eligibility for the NPP. It will include those who have already completed T-DXd treatment under the NPP, as well as patients whose T-DXd treatment remains ongoing.
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Real-World Time-to-Treatment Discontinuation In Participants Treated With Trastuzumab Deruxtecan (T-DXd) | From the time from T-DXd initiation to the date of T-DXd discontinuation, up to 14 months
  Real-world time-to-treatment discontinuation (rwTTD) is defined as the time from trastuzumab deruxtecan initiation to discontinuation for any reason in patients with advanced/metastatic HER2+ breast cancer in a real-world clinical setting.

SECONDARY OUTCOMES:
Type of Prior Targeted HER2-targeted Treatments In Participants Treated With Trastuzumab Deruxtecan (T-DXd) | Prior to time of T-DXd initiation
Number of Participants Who Discontinued Trastuzumab Deruxtecan (T-DXd) In Participants Treated With T-DXd | From the time from T-DXd initiation to the date of T-DXd discontinuation, up to 14 months
Number of Participants With Treatment-emergent Adverse Events In Participants Treated With Trastuzumab Deruxtecan (T-DXd) | From the time from T-DXd initiation to the date of T-DXd discontinuation, up to 14 months
Number of Participants Who Received Prophylaxis Treatment In Participants Treated With Trastuzumab Deruxtecan (T-DXd) | Prior to time of T-DXd initiation
  Patients who received prophylaxis treatment for nausea and/or vomiting will be reported.
Real World Progression-free Survival In Participants Treated With Trastuzumab Deruxtecan (T-DXd) | From the time of T-DXd initiation to the date of T-DXd discontinuation, withdrawal, or disease progression, up to 14 months
  Real world progression-free survival (rwPFS) is defined as the time from T-DXd initiation to the earliest of death or progression.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (21):
- Ireland (2):
  - St. Vincent's Private Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
- Italy (7):
  - Breast Center Humanitas Cancer Center IRCCS Istituto Clinico Humanitas, Rozzano, Milano
  - Centro di riferimento Oncologico (CRO), National Cancer Institute, Aviano, Pordenone
  - National Cancer Instutute 'Fondazione Pascale, Naples
  - Institute Oncology Veneto, Padua
  - Universita Campus Bio-Medico Di Roma, Rome
  - Policlinico Umberto I Di Roma, Rome
  - Fondazione Policlinico Univeritario Agostino Gemeli, Rome
- Spain (12):
  - Hospital General Universitario De Alicante, Alicante
  - Hospital Del Mar, Barcelona
  - Hospital Quiron Salud Barcelona, Barcelona
  - Hospital Val d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - ICO Girona, Girona
  - Hospital Universitario de Jaen, Jaén
  - Hospital Clínico San Carlos, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Fundacion Instituto Valenciano de Oncologia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saura C, Wildiers H, Bianchini G, Garcia-Saenz JA, Allignol A, Logue A, Lucerna M, Stamenitis S, De Laurentiis M. European experience of patients with HER2-positive advanced/metastatic breast cancer accessing trastuzumab deruxtecan through a named patient program: the EUROPA T-DXd study. Front Oncol. 2025 Oct 14;15:1650981. doi: 10.3389/fonc.2025.1650981. eCollection 2025. PMID 41164130